CLINICAL TRIAL: NCT06706934
Title: Search for Phenotype-modifying Genes in Patients With Intellectual Disabilities GWAS-2DI.
Brief Title: Search for Phenotype-modifying Genes in Patients With Intellectual Disabilities.
Acronym: GWAS-2DI
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2024 75
Record Dates: First submitted 2024-11-22; First posted 2024-11-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-11

CONDITIONS: Intellectual Disability
Keywords: Intellectual Disability; epistatic interaction
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients group with intellectual disability
- Control: Control group without intellectual disability

SUMMARY:
Each form of intellectual disability under study is a rare disease in its own right, and it is therefore difficult to study the variability of its expression. It therefore appears necessary to study large series of patients with intellectual disabilities. The objective is to identify variants in phenotype-modifying genes in patients with intellectual disability.

DETAILED DESCRIPTION:
Thanks to the contribution of NGS analyses (exome and genome analysis), the rate of etiological diagnosis in intellectual disability is currently approaching 42% in some meta-analyses. At Bordeaux University Hospital, since 2017, 700 patients have been sequenced for intellectual disability, with a diagnostic rate of 33%.

In genetics, epistasis refers to the interaction between two or more genes. As part of its previous work, BIONOMEEX has developed an algorithm called GWAS-2D (genome wide association study 2 dimension) which makes it possible to observe, from a large number of samples and for a given phenotype, the relationships existing between two loci on the genome.

The GWAS-2DI project involves the reanalysis of exome sequencing data from patients with intellectual disabilities at Bordeaux University Hospital, using a GWAS-2D algorithm developed by BIONOMEEX to search for phenotype-modifying genes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Intellectual Disability or related but not affected by them
* Major or minor with autorisation of legal representative
* Exome sequencing in Bordeaux University Hospital between 2018 and 2024

Exclusion Criteria:

* Refusal to participate in research protocols
* Refusal to participate expressed following receipt of information letter.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with intellectual disabilities or related but not affected by them
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Variants in phenotype-modifying genes | Inclusion visit
  Identifying variants in phenotype-modifying genes in patients with intellectual disability.

SECONDARY OUTCOMES:
Phenotypic traits | Inclusion visit
  Correlation phenotypic traits with additional diagnostic variants

CONTACTS AND LOCATIONS:
Overall Officials: Vincent MICHAUD, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Chu de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No